CLINICAL TRIAL: NCT05258890
Title: TEAMS-BP (The Enhancement of Social Networks to Augment Management of Stroke-Blood Pressure): A Randomized Control Trial
Brief Title: TEAMS-BP (The Enhancement of Social Networks to Augment Management of Stroke-Blood Pressure)
Acronym: TEAMS-BP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment and poor retention despite several efforts to overcome these hurdles
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amar Dhand, MD DPhil, Associate Professor of Neurology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022P000444; 5P30AG064199-03 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute Ischemic; Hypertension
Keywords: Social Networks
MeSH Terms: conditions — Ischemic Stroke; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Network Counseling (Experimental): The index patient and influential social network members will meet via Zoom 3 times over the course of 3 months with a clinical research nurse for teamwork counseling and blood pressure education.
  Interventions: Other: Social Network Group Counseling
- Individual Counseling (Active Comparator): The index patient will meet via Zoom 3 times over the course of 3 months with a clinical research nurse for blood pressure education.
  Interventions: Other: Individual Counseling

INTERVENTIONS:
Other: Social Network Group Counseling — Researchers will identify the influential network members based on their network position, driving distance from the patient, speaking frequency, and whether they have high blood pressure. The index patient and social network members will meet with the study nurse on weeks 2, 6, and 12 after initial enrollment. The study nurse will begin the social network counseling session in which she will provide counseling on teamwork and blood pressure control. The teamwork specific topics will include how networks can work together as a team, communication tips for engaging with one another, spreading positive messages, and establishing the roles and responsibilities of each network team member. The blood pressure control specific topics will include the basics of blood pressure, taking and adjusting medications, monitoring blood pressure, reducing salt, and being physically active. Patient and social network members will receive text messages every week in the weeks between sessions.
  Arms: Social Network Counseling
Other: Individual Counseling — The index patient will meet individually with the study nurse on weeks 2, 6, and 12 after initial enrollment. The nurse will provide counseling on the basics of blood pressure, taking and adjusting medications, monitoring blood pressure, reducing salt, and being physically active. The patient will receive text messages every week in the weeks between sessions.
  Arms: Individual Counseling

SUMMARY:
This study aims to compare the efficacy of a social network intervention versus individual hypertension counseling to improve blood pressure control after stroke. The investigators hope to understand whether the involvement of family, friends and other members of individual's social network can help achieve better blood pressure after experiencing a stroke. Participants will be stratified to two groups according to network size (<5 vs 5 or more) and randomized to receive individual hypertension counseling (control) or the social network intervention. The primary outcome of the study will be the absolute reduction in systolic blood pressure at 3 months follow-up. The secondary outcomes will be attainment of a post-stroke hypertension treatment goal and patient-reported physical function.

ELIGIBILITY:
Inclusion Criteria:

1. First acute ischemic stroke defined clinically with support from imaging if necessary
2. 21 years of age or older
3. Within 14 days after stroke
4. History of hypertension or has been newly prescribed blood pressure medications during index admission

Exclusion Criteria:

1. Prior ischemic or hemorrhagic stroke
2. NIHSS > 21
3. Significant aphasia (Score>1 on the language section of the NIHSS)
4. Medical conditions for which death is likely within 6 months
5. Does not have capacity to consent for the project or participate in survey interview
6. Diagnosis of dementia
7. Patient has no phone or incapable of using text messages
8. Patient has opted out of participating in research noted within MGB Epic EHR system

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Dhand, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhand A, Crum K, Hanken KE, Bhatkhande G, Luo M, Corbin IM, Usmanov G, Rothfeld-Wehrwein Z, Dhongade V, Lin D, Slocum C, Haff N, Choudhry NK. Social network intervention to improve blood pressure control after stroke: The TEAMS-BP randomized clinical trial. Soc Sci Med. 2025 Sep;380:118231. doi: 10.1016/j.socscimed.2025.118231. Epub 2025 May 21. PMID 40414088

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 47 patients enrolled, but 2 patients withdrew prior to randomization. Social network members were only enrolled in the social network counseling arm. All consented patients' social network members were collected in the baseline questionnaire, prior to randomization. For patients who were randomized to individual counseling (n=21), network members were not enrolled. For patients who were randomized to social network counseling (n=24), network members were enrolled (n=17).
Period: Overall Study
Arm/Group | Social Network Counseling | Individual Counseling
Started | 41 | 21
Index Patients Who Started | 24 | 21
Social Network Members Who Started Members | 17 | 0 (Per the protocol, social network members were not enrolled for patients randomized to this arm.)
Completed | 19 (8 patients and 11 social networks members completed the study.) | 11
Not Completed | 22 | 10
Not completed — Patient withdrawal | 6 | 7
Not completed — Patient lost to follow-up | 10 | 3
Not completed — Social network member withdrawal | 1 | 0
Not completed — Social network member lost to follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were not collected for social network members.
Groups:
- Social Network Counseling - Patients Only: The index patient and influential social network members will meet via Zoom 3 times over the course of 3 months with a clinical research nurse for teamwork counseling and blood pressure education.
  Social Network Group Counseling: Researchers will identify the influential network members based on their network position, driving distance from the patient, speaking frequency, and whether they have high blood pressure. The index patient and social network members will meet with the study nurse on weeks 2, 6, and 12 after initial enrollment. The study nurse will begin the social network counseling session in which she will provide counseling on teamwork and blood pressure control. The teamwork specific topics will include how networks can work together as a team, communication tips for engaging with one another, spreading positive messages, and establishing the roles and responsibilities of each network team member. The blood pressure control specific topics will include the basics of blood pressure, taking and adjusting medications, monitoring blood pressure, reducing salt, and being physically active. Patient and social network members will receive text messages every week in the weeks between sessions.
- Individual Counseling - Patients Only: The index patient will meet via Zoom 3 times over the course of 3 months with a clinical research nurse for blood pressure education.
  Individual Counseling: The index patient will meet individually with the study nurse on weeks 2, 6, and 12 after initial enrollment. The nurse will provide counseling on the basics of blood pressure, taking and adjusting medications, monitoring blood pressure, reducing salt, and being physically active. The patient will receive text messages every week in the weeks between sessions.
- Total: Total of all reporting groups
Arm/Group | Social Network Counseling - Patients Only | Individual Counseling - Patients Only | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.41 (13.46) | 70.71 (10.41) | 67.36 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 15 | 12 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 7 | 3 | 10
  White | 15 | 16 | 31
  Asian | 1 | 0 | 1
  Other | 1 | 2 | 3
Ethnicity [Count of Participants; unit: Participants]
  Hisapnic/Latino | 1 | 2 | 3
  Not Hispanic/Latino | 22 | 18 | 40
  Unknown | 1 | 1 | 2
Baseline Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 135.32 (21.74) | 145.81 (21.05) | 140.44 (21.55)
Education level [Count of Participants; unit: Participants]
  Some high school or less | 2 | 0 | 2
  High school graduate | 4 | 7 | 11
  Some college | 4 | 5 | 9
  Associate degree | 2 | 2 | 4
  Bachelor's degree | 5 | 4 | 9
  Graduate degree | 6 | 3 | 9
  Prefer not to answer | 1 | 0 | 1
Employment status [Count of Participants; unit: Participants]
  Retired | 9 | 9 | 18
  Employed | 9 | 7 | 16
  Self-employed | 2 | 4 | 6
  Other | 4 | 1 | 5
Marital Status [Count of Participants; unit: Participants]
  Not married | 13 | 11 | 24
  Married | 11 | 10 | 21
Social network size [Mean (Standard Deviation); unit: Network members] | 4.92 (3.24) | 5.86 (4.45) | 5.36 (3.84)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure for Patient-Subjects
Description: Blood pressure was not collected for social network members.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Social Network Counseling | Individual Counseling
Number analyzed (Participants) | 24 | 21
mmHg | -10.82 (5.08) | -5.31 (6.10)

2. Secondary Outcome: Achievement of Post-stroke Hypertension Treatment Goal for Patient-Subjects
Description: This was evaluated as achieving a blood pressure of <130/80 mmHg. Blood pressure was not collected for social network members.
Time Frame: 3 months
Population: This was only assessed for those patient subjects who completed the 3-month follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Social Network Counseling | Individual Counseling
Number analyzed (Participants) | 8 | 11
Participants | 5 | 3

3. Secondary Outcome: Patient Reported Physical Function for Patient-Subjets
Description: This was evaluated for patient-subjects only (not collected for social network subjects), using the validated Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) scale.
  For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
  The T-score is provided with an error term (Standard Error or SE). The Standard Error is a statistical measure of variance and represents the "margin of error" for the T-score.
  A higher PROMIS T-score represents better physical function. A T-score of 60 indicates one SD better than the average physical function for the United States general population.
Time Frame: 3 months
Population: This was only assessed for those patient-subjects who completed the 3-month follow-up period.
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Social Network Counseling | Individual Counseling
Number analyzed (Participants) | 8 | 11
T-score on a scale | 37.48 (12.88) | 45.25 (12.20)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through the end of the 3 month study follow-up period.
Description: Adverse events were only collected for patient-subjects.
  The social network members were enrolled as support for the enrolled index patient, and therefore, were not at risk of study-related adverse events since there was not an intervention targeting the social network members.
Arm/Group | Social Network Counseling | Individual Counseling
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/24 | 2/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Social Network Counseling (N=24) | Individual Counseling (N=21)
Acute/subacute ischemic stroke (Nervous system disorders) | 0 | 2
Planned surgery of carotid artery (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT05258890/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT05258890/ICF_000.pdf